CLINICAL TRIAL: NCT01171053
Title: Internet-delivered Exposure and Mindfulness Based Therapy for Irritable Bowel Syndrome - A Randomized Controlled Trial
Brief Title: Internet-delivered CBT for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Nils Lindefors, Psykiatri Sydväst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBS-S
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Cognitive behavior therapy; Internet; Cost-effectiveness; Irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention control (Placebo Comparator): Weekly support from therapist without CBT-interventions
  Interventions: Behavioral: Therapist support
- Internet CBT (Experimental): Internet-delivered cognitive behavioral therapy with therapist support
  Interventions: Behavioral: Internet-delivered CBT

INTERVENTIONS:
Behavioral: Internet-delivered CBT — Internet-delivered cognitive behavioral therapy with therapist support.
  Arms: Internet CBT
Behavioral: Therapist support — Weekly therapist support without CBT-interventions
  Arms: Attention control

SUMMARY:
The aim of this study is to investigate the efficacy of a 10 week Internet-delivered CBT treatment for patients diagnosed with IBS. The patients' work with the treatment and is supported through online contact with a therapist.

Approximately 86 patients will be included in the study and randomized to either condition.

All included patients are assessed one week before the treatment starts. After 10 weeks (post treatment). Follow-up assessments are conducted at 3 and 12 months follow-up after treatment.

Patients in treatment condition are hypothesized to experience significant reduction IBS symptoms, societal costs and quality of life compared to patients on waiting list.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBS given by physician
* At screening fulfilling Rome III-criteria for IBS

Exclusion Criteria:

* Severe depression
* Suicidal ideation
* Presence of unexplained IBS alarm symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | One week before the treatment starts
  Gastrointestinal Symptom rating scale (GSRS)
Gastrointestinal symptoms | 10 weeks after the treatment started
  Gastrointestinal Symptom rating scale (GSRS)
Gastrointestinal symptoms | 3 months after the treatment ended
  Gastrointestinal Symptom rating scale (GSRS)
Gastrointestinal symptoms | One year after the treatment ended
  Gastrointestinal Symptom rating scale (GSRS)

SECONDARY OUTCOMES:
Health economic data | One week before the treatment starts
  "Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry". In this questionnaire, patients register their monthly health care consumption (e.g. GP visits) as well as time spent in informal health enhancing activities (e.g. self-help groups and informal care from friends). In addition, work loss and work cutback both at work and in the domestic realm is measured.
Health economic data | 10 weeks after the treatment started
  "Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry". In this questionnaire, patients register their monthly health care consumption (e.g. GP visits) as well as time spent in informal health enhancing activities (e.g. self-help groups and informal care from friends). In addition, work loss and work cutback both at work and in the domestic realm is measured.
Health economic data | 3 months after the treatment ended
  "Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry". In this questionnaire, patients register their monthly health care consumption (e.g. GP visits) as well as time spent in informal health enhancing activities (e.g. self-help groups and informal care from friends). In addition, work loss and work cutback both at work and in the domestic realm is measured.
Health economic data | One year after the treatment ended
  "Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry". In this questionnaire, patients register their monthly health care consumption (e.g. GP visits) as well as time spent in informal health enhancing activities (e.g. self-help groups and informal care from friends). In addition, work loss and work cutback both at work and in the domestic realm is measured.
Quality of life | One week before the treatment starts
  The Irritable Bowel Syndrome Quality of Life Instrument
Quality of life | 10 weeks after the treatment started
  The Irritable Bowel Syndrome Quality of Life Instrument
Quality of life | 3 months after the treatment ended
  The Irritable Bowel Syndrome Quality of Life Instrument
Quality of life | One year after the treatment ended
  The Irritable Bowel Syndrome Quality of Life Instrument
Gastrointestinal symptom-specific anxiety | One week before the treatment starts
  Visceral Sensitivity Index
Gastrointestinal symptom-specific anxiety | 10 weeks after the treatment started
  Visceral Sensitivity Index
Gastrointestinal symptom-specific anxiety | 3 months after the treatment ended
  Visceral Sensitivity Index
Gastrointestinal symptom-specific anxiety | One year after the treatment ended
  Visceral Sensitivity Index
Depressive symptoms | One week before the treatment starts
  The Montgomery Åsberg Depression Rating Scale
Depressive symptoms | 10 weeks after the treatment started
  The Montgomery Åsberg Depression Rating Scale
Depressive symptoms | 3 months after the treatment ended
  The Montgomery Åsberg Depression Rating Scale
Depressive symptoms | One year after the treatment ended
  The Montgomery Åsberg Depression Rating Scale
Functional impairments in work, social and family life | One week before the treatment starts
  Sheenan Disability Scale (DSD)
Functional impairments in work, social and family life | 10 weeks after the treatment started
  Sheenan Disability Scale (DSD)
Functional impairments in work, social and family life | 3 months after the treatment ended
  Sheenan Disability Scale (DSD)
Functional impairments in work, social and family life | One year after the treatment ended
  Sheenan Disability Scale (DSD)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Lindefors, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykatrienheten, M46, Psykiatri sydväst, Stockholm, Sweden

REFERENCES:
- [Result] Ljotsson B, Falk L, Vesterlund AW, Hedman E, Lindfors P, Ruck C, Hursti T, Andreewitch S, Jansson L, Lindefors N, Andersson G. Internet-delivered exposure and mindfulness based therapy for irritable bowel syndrome--a randomized controlled trial. Behav Res Ther. 2010 Jun;48(6):531-9. doi: 10.1016/j.brat.2010.03.003. Epub 2010 Mar 16. PMID 20362976